CLINICAL TRIAL: NCT05044013
Title: Training in mHealth Prevention With MSM
Brief Title: Testing of the Smartphone App to Enhance HIV Prevention Cascade Among Malaysian MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other); Yale University (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01DA051346 (NIH)
Record Dates: First submitted 2021-08-25; First posted 2021-09-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HIV Prevention Program
Keywords: mobile application; PrEP; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JomPrEP App Group (Experimental): Participants in the JomPrEP group will be provided with full app access and will be encouraged to use all features of the app.
  Interventions: Other: Full access to JomPrEP app
- Control Group (Active Comparator): Participants in the control group will receive the JomPrEP app with major intervention features inactivated.
  Interventions: Other: inactivated JomPrEP app

INTERVENTIONS:
Other: Full access to JomPrEP app — All participants will receive the JomPrEP app with access to all of its features which include: customizable page (using avatars and pseudonyms); visual dashboard (track and visualize progress); HIV testing plan (create plan for HIV testing, order self-testing kits, testing site locator); PrEP Care Plan (PrEPxpress, automated reminders for follow-up care, labs, delivery); chat function and discussion forum; tailored messages and reminders; assessment center (weekly assessment on adherence to PrEP, HIV risk, mood); knowledge center (resources on HIV testing and PrEP); Mental health support (screen for P/SUD, counseling feedback, referral to support services); Integration of provider locator (provides users with a GPS enabled map for PrEP and mental health support providers in Malaysia) and Gamification (offers extrinsic motivation by rewarding points/milestones for doing activities within the app). Participants can also contact the RA using the chat function for support.
  Arms: JomPrEP App Group
Other: inactivated JomPrEP app — Only information and resources for PrEP services will be available along with access to risk assessment tools.
  Arms: Control Group

SUMMARY:
The investigators will conduct a pilot RCT to evaluate the feasibility and acceptability of the JomPrEP app and examine its preliminary efficacy in improving PrEP cascade compared with the control group.

DETAILED DESCRIPTION:
mHealth is a promising and cost-effective strategy to reach stigmatized and hard-to-reach populations and link them to care. Leveraging mHealth reduces individuals' discomfort and distrust of disclosing risk behaviors to providers, providers' low cultural competency for working with individuals of diverse sexual identities, and bypasses barriers to care for marginalized populations, - all features crucial for HIV prevention in MSM in Malaysia. Results from the investigators' studies show Malaysian MSM often do not get HIV tested or initiate PrEP. Mixed methods suggest MSM want these services but prefer a streamlined system to access them that reduces interaction with clinicians where disclosure and perceived judgment occurs. mHealth may overcome these barriers by facilitating prevention services delivery and health decision-making in a confidential, less-stigmatizing, and convenient manner. Overall smartphone growth in Malaysia (63% in 2015 to 89% in 2017), and the investigators' parallel work with MSM indicates that nearly all (>97%) MSM own a smartphone. Findings from qualitative interviews with MSM further indicate preferences for interfacing with 'apps' rather than health professionals as well as local stakeholders indicating strong interest in using such platform to deliver HIV prevention services align with developing culturally tailored mHealth strategies and to engage MSM in virtual communication with providers - all embedded within one app.

To the investigators' knowledge however, no mHealth intervention has been developed to improve access to HIV prevention services in Malaysia. The investigators, therefore, propose to pilot test their new clinic-affiliated app (JomPrEP) to promote HIV testing and PrEP uptake in Malaysian MSM. They will conduct a pilot RCT to evaluate the feasibility and acceptability of the JomPrEP app and examine its preliminary efficacy in improving PrEP cascade compared with the control group.

The investigators will enroll 90 participants who will be randomized (1:1) to receive either the JomPrEP app or the control group and assessed at 3- and 6-months. Randomization will be stratified by ATS use (16% to 24%) and age. They will conduct exit interviews with participants and clinical staff to examine the barriers and facilitators to the app and obtain feedback to further optimize the app.

ELIGIBILITY:
Inclusion Criteria: MSM

* HIV-negative MSM
* Age more than or equal to 18
* Cis-gender men
* Condomless sex in the last 30 days
* Own a smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender men
Enrollment: 90 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the JomPrEP app using percentages of individuals screened | 6 months
  The investigators will use the percentage of individuals screened to determine the feasibility of the JomPrEP app
Feasibility of the JomPrEP app using percentages of individuals eligible | 6 months
  The investigators will use the percentage of individuals eligible to determine the feasibility of the JomPrEP app
Feasibility of the JomPrEP app using percentages of individuals enrolled | 6 months
  The investigators will use the percentage of individuals enrolled to determine the feasibility of the JomPrEP app
Feasibility of the JomPrEP app using percentages of individuals retained | 6 months
  The investigators will use the percentage of individuals retained to determine the feasibility of the JomPrEP app
Feasibility of the JomPrEP app using the percentage of participants that accessed the app | 6 months
  The investigators will determine the percentage of participants that accessed the app, with ≥60% of participants accessing app as lower threshold. The higher the percentage, the higher the feasibility.
Acceptability of the JomPrEP app based on the subjective usability measure | 6 months
  Acceptability will be based on descriptive statistics from the subjective usability measure, with a target mean score of ≥ 50. The higher the score, the higher the acceptability. Minimum score for the scale is 0, highest is 100.
Acceptability of the JomPrEP app based on perceived usefulness of participants assessed in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes specific areas of perceived usefulness of the app.
Acceptability of the JomPrEP app based on barriers and facilitators identifies by participants in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes barriers and facilitators.
Acceptability of the JomPrEP app based on usability concerns identified by participants in qualitative interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes usability concerns.
Acceptability of the JomPrEP app based on refinement feedback identified by participants in qualitative data interviews | 6 months
  Acceptability will be based on analysis of qualitative data which includes refinement needed to maximize future implementation.

SECONDARY OUTCOMES:
Preliminary Efficacy of the JomPrEP app through dried blood spot testing as PrEP adherence measure | 3 months
  The investigators will measure PrEP adherence (using dried blood spots) at 3 months. DBS will quantify tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in RBC.
Preliminary Efficacy of the JomPrEP app through dried blood spot testing as PrEP adherence measure | 6 months
  The investigators will measure PrEP adherence (using dried blood spots) at 6 months. DBS will quantify tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in RBC
Preliminary Efficacy of the JomPrEP app using the visual analog scale (VAS) to measure PrEP adherence | 3 months
  The investigators will measure PrEP adherence using the visual analogue scale at 3 months.
Preliminary Efficacy of the JomPrEP app using the visual analog scale (VAS) to measure PrEP adherence | 6 months
  The investigators will measure PrEP adherence using the visual analogue scale at 6 months.
Preliminary Efficacy of the JomPrEP app using proportion of participants who persist on PrEP | 6 months
  Preliminary Efficacy of the app will be calculated using the proportion of participants who persist on PrEP. Persistence on PrEP is measured on the app when completing PrEP care.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Shrestha, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Centre of Excellence For Research in AIDS (CERiA), Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Van Tieu H, Koblin BA. HIV, alcohol, and noninjection drug use. Curr Opin HIV AIDS. 2009 Jul;4(4):314-8. doi: 10.1097/COH.0b013e32832aa902. PMID 19532070
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Guadamuz TE, Cheung DH, Wei C, Koe S, Lim SH. Young, Online and in the Dark: Scaling Up HIV Testing among MSM in ASEAN. PLoS One. 2015 May 14;10(5):e0126658. doi: 10.1371/journal.pone.0126658. eCollection 2015. PMID 25973907
- [Background] Giordano TP, Guzman D, Clark R, Charlebois ED, Bangsberg DR. Measuring adherence to antiretroviral therapy in a diverse population using a visual analogue scale. HIV Clin Trials. 2004 Mar-Apr;5(2):74-9. doi: 10.1310/JFXH-G3X2-EYM6-D6UG. PMID 15116282
- [Background] Grant RM, Anderson PL, McMahan V, Liu A, Amico KR, Mehrotra M, Hosek S, Mosquera C, Casapia M, Montoya O, Buchbinder S, Veloso VG, Mayer K, Chariyalertsak S, Bekker LG, Kallas EG, Schechter M, Guanira J, Bushman L, Burns DN, Rooney JF, Glidden DV; iPrEx study team. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. Lancet Infect Dis. 2014 Sep;14(9):820-9. doi: 10.1016/S1473-3099(14)70847-3. Epub 2014 Jul 22. PMID 25065857
- [Background] Castillo-Mancilla JR, Zheng JH, Rower JE, Meditz A, Gardner EM, Predhomme J, Fernandez C, Langness J, Kiser JJ, Bushman LR, Anderson PL. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. AIDS Res Hum Retroviruses. 2013 Feb;29(2):384-90. doi: 10.1089/AID.2012.0089. Epub 2012 Oct 10. PMID 22935078
- [Background] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401
- [Background] Zheng JH, Rower C, McAllister K, Castillo-Mancilla J, Klein B, Meditz A, Guida LA, Kiser JJ, Bushman LR, Anderson PL. Application of an intracellular assay for determination of tenofovir-diphosphate and emtricitabine-triphosphate from erythrocytes using dried blood spots. J Pharm Biomed Anal. 2016 Apr 15;122:16-20. doi: 10.1016/j.jpba.2016.01.038. Epub 2016 Jan 21. PMID 26829517
- See also: Determining What Individual SUS Scores Mean: Adding an Adjective Rating Scale by Aaron Bangor, PhD, CHFP, Philip Kortum, PhD, James Miller, PhD — https://uxpajournal.org/determining-what-individual-sus-scores-mean-adding-an-adjective-rating-scale/
- See also: Transforming Qualitative Information Thematic Analysis and Code Development. By Richard E. Boyatzis — https://us.sagepub.com/en-us/nam/transforming-qualitative-information/book7714
- See also: Handbook of data analysis. By Roberto P. Franzosi. — https://dokumen.pub/the-handbook-of-data-analysis-7-1nbsped-1848601166-978-1-84860-116-1.html